CLINICAL TRIAL: NCT05738681
Title: Efficacy of N-acetylcysteine to Prevent Anti-tuberculosis Drug-induced Liver Injury: A Randomized Controlled Trial
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Watcharasak Chotiyaputta, Associate professor, Faculty of Medicine, Siriraj Hospital Affiliation: Mahidol University, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Si 1052/2020
Record Dates: First submitted 2022-07-11; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Tuberculosis; Drug Induced Liver Injury; Hepatitis
Keywords: Tuberculosis; DILI; Anti tuberculosis
MeSH Terms: conditions — Tuberculosis; Chemical and Drug Induced Liver Injury; Hepatitis | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Tuberculosis patients who had standard regimen treatment, non-HIV, no severe co-morbidity, no chronic hepatitis B or C were randomized to using NAC-long 1,200 mg/day for 8 weeks (NAC long group) or using anti-TB alone (non-NAC group). Genetic test, CBC, Cr, coagulogram were assessed at baseline. LFT were assessed at baseline, 2 weeks, 8 weeks and 24 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NAC group (Experimental): Tuberculosis patients who had standard regimen treatment, non-HIV, no severe co-morbidity, no chronic hepatitis B or C using NAC-long 1,200 mg/day for 8 weeks (NAC long group). Genetic test (acetylator status of NAT2), CBC, Cr, coagulogram were assessed at baseline. LFT were assessed at baseline, 2 weeks, 8 weeks and 24 weeks.
  Interventions: Drug: N acetyl cysteine
- Non-NAC group (No Intervention): Tuberculosis patients who had standard regimen treatment, non-HIV, no severe co-morbidity, no chronic hepatitis B or C were using anti-TB alone (non-NAC group). Genetic test (Acetylator status of NAT2), CBC, Cr, coagulogram were assessed at baseline. LFT were assessed at baseline, 2 weeks, 8 weeks and 24 weeks.

INTERVENTIONS:
Drug: N acetyl cysteine — N acetyl cysteine 1,200 mg/day for 8 weeks in NAC group
  Other Names: Standard anti TB drug regimen
  Arms: NAC group

SUMMARY:
To determine the efficacy of NAC to prevent clinically significant anti-TB drugs induced liver injury (AT-DILI).

DETAILED DESCRIPTION:
Tuberculosis is one of the most important infectious diseases and treatment related hepatitis from anti-TB drug was observed for 5-28%. Slow acetylator status in the N-acetyltransferase 2 (NAT2) genotype is a significant risk factor of anti-tuberculosis drug-induced liver injury (AT-DILI). We assessed the effect of N-acetylcysteine to prevent hepatitis from anti-TB drug in Thai population.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed TB
* Received standard dose of anti-TB drugs regimen (National Tuberculosis Control Programme guideline Thailand 2018)
* Aged ≥18 years
* Informed consent

Exclusion Criteria:

* Previous TB infection or MDR TB
* TB liver
* Allergy to NAC
* Abnormal baseline LFT
* (AST or ALT>2.5 times UNL, ALP> 2 times UNL, TB> 1.5 mg/dl)
* Chronic hepatitis B, C infection
* Decompensated cirrhosis
* HIV infection
* Active malignancy
* Pregnancy or lactation
* Severe co-morbidity i.e. severe heart diseases, severe lung diseases, ESRD

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hepatitis at 8 weeks | 8 weeks
  To study efficacy of NAC to prevent anti-TB drug induced liver injury. Outcome was measured events of hepatitis occurred at 8 weeks, compared between NAC versus controlled group, presented by total number and percent.
  Significant hepatitis was defined as elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than 5 times of baseline levels.

SECONDARY OUTCOMES:
Prevalence of hepatitis among NAT2 slow acetylator patients | 8 weeks
  To study efficacy of NAC to prevent anti-TB drug induced liver injury among NAT2 slow acetylator patients.
  Outcome was measured events of hepatitis occurred at 8 weeks among NAT2 slow acetylator patients compared between NAC versus controlled group, presented by total number and percent.
  Significant hepatitis was defined as elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than 5 times of baseline levels.

OTHER OUTCOMES:
Prevalence of hepatitis at 2 weeks | 2 weeks
  Outcome was measured events of hepatitis occurred at 2 weeks, compared between NAC versus controlled group, presented by total number and percent.
  Significant hepatitis was defined as elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than 5 times of baseline levels.
Prevalence of hepatitis at 24 weeks | 24 weeks
  Outcome was measured events of hepatitis occurred at 24 weeks, compared between NAC versus controlled group, presented by total number and percent.
  Significant hepatitis was defined as elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than 5 times of baseline levels.

CONTACTS AND LOCATIONS:
Overall Officials: Supot Nimanong, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Patient data may be secure and not sharing